CLINICAL TRIAL: NCT06092411
Title: Effects of Cognitive Behavioural Therapy and Bright Light Therapy in Youth With Unipolar Depression and Evening Chronotype: An Assessor-blind Parallel-group Randomised Controlled Trial
Brief Title: Effects of CBT and BLT in Youth With Unipolar Depression and Evening Chronotype
Acronym: DELAY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA220381
Record Dates: First submitted 2023-09-19; First posted 2023-10-23 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Depression, Unipolar; Eveningness
Keywords: Depression; Eveningness; Adolescents; Bright Light Therapy; Cognitive Behavioural Therapy
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Cognitive Behavioral Therapy; Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT for Depression + Bright Light Therapy (CBTD+BLT) (Experimental): N = 54
  Interventions: Behavioral: Cognitive Behavioural Therapy for Depression; Device: Bright Light Therapy
- CBT for Depression + Placebo Light (CBTD-BLT) (Active Comparator): N = 54
  Interventions: Behavioral: Cognitive Behavioural Therapy for Depression
- Waitlist Control (WL) (No Intervention): N = 54

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Depression — Consists of 8 weekly sessions (group-based, 90-min, 4-6 adolescents in each group). The intervention focuses on addressing depression, with the components such as psycho-education on depression, self-monitoring, behavioural activation, and cognitive restructuring (addressing negative and irrational thoughts often associated with depression in adolescents), relaxation techniques, and relapse prevention.
  Arms: CBT for Depression + Bright Light Therapy (CBTD+BLT); CBT for Depression + Placebo Light (CBTD-BLT)
Device: Bright Light Therapy — Participants will undergo daily morning light therapy by wearing a validated portable light emitting device (i.e., Re-Timers: https://www.re-timer.com/) at home for 30 minutes. Participants will receive bright blue-green light (500 nm, 506 lux).
  Arms: CBT for Depression + Bright Light Therapy (CBTD+BLT)

SUMMARY:
The goal of this prospective randomised controlled trial is to examine the effects of cognitive behavioural therapy and bright light therapy in youths with unipolar depression and evening chronotype. The main questions it aims to answer are:

1. What is the efficacy of CBT-D and CBT-D plus bright light therapy in reducing depression severity in adolescents with depression and eveningness?
2. What are the effects of CBT-D and CBT-D plus bright light therapy on the subjective and objective sleep and circadian measures, as well as the quality of life, daytime symptoms, and functioning (e.g., sleepiness, fatigue)?

Participants will participate in 8 weekly group sessions of CBT-D intervention based on the well-established CBT elements for treating depression. Concurrently participants will also be asked to wear a portable light device at home for 30 minutes daily for seven weeks, starting from the second week of the group intervention. Participants in the CBT-D only group will receive a placebo light via the device, whereas participants in the CBT-D plus light therapy group will receive the active bright light via the device.

DETAILED DESCRIPTION:
Adolescence is a vulnerable period often linked to the emergence of emotional and behavioural difficulties, particularly major depressive disorder (MDD). It is also associated with a gradual change of circadian rhythm characterised by an intrinsic phase delay with an increased evening preference linked to pubertal development. The optimal treatment for youth depression remains controversial. CBT for depression (CBT-D) is one of the most extensively tested psychological treatments for managing mild to moderate depression. Nonetheless, well-designed randomised controlled trials (RCTs) of CBT-D conducted in young people were limited, and the existing research showed that more than 60% of youth did not respond to psychological treatments. Therefore, improving the current model of care and outcomes in youth with depression is imperative, yet rigorous controlled trials of the treatment for youth depression remain limited. In addition, despite the close interplay between circadian disruption and mood problems, little is known as to whether the adjunctive circadian-focused intervention could potentially enhance the treatment outcome of adolescent depression, especially in those with circadian vulnerability (eveningness).

The study is a randomised controlled trial that examines the effects of cognitive behavioural therapy and bright light therapy in youth with unipolar depression and evening chronotype. Eligible participants will be randomised to one of the following groups: CBT-D plus bright light therapy (CBTD+BLT), CBT for depression only (CBTD-BLT), or waiting list control (WL) using an automated online system. For both treatment groups, the intervention will consist of 8 weekly group sessions (90-min, 4-6 adolescents in each group) of CBT-D delivered in the afternoon/evening after school within a 10-week window. The intervention is structured and based on the well-established CBT elements for treating depression, which combines cognitive and behavioural strategies targeting the common difficulties and problems encountered by depressed adolescents. Participants in both treatment groups will also be introduced to the daily light-based intervention by wearing a portable light device (Re-timers) at home for 30 minutes daily for seven weeks, starting from the second week of the group intervention. Participants in the CBTD-BLT group will receive a placebo light intervention, where they will be exposed to dim red light (50 lux), whereas participants in the CBT-D plus light therapy group will receive the active light treatment. All participants initially randomised to the WL condition will be offered treatment opportunities at the end of the WL period.

The primary aim of the study is to test the efficacy of CBT-D and CBT-D plus bright light therapy in reducing depression severity in adolescents with depression and eveningness when compared with the waiting list control. The secondary aim of the study is to examine the effects of CBT-D and CBT-D plus bright light therapy on the subjective and objective sleep and circadian measures, as well as the measures of quality of life, daytime symptoms and functioning (e.g., sleepiness, fatigue).

ELIGIBILITY:
Inclusion Criteria:

1. Chinese aged 12-20 years old.
2. Written informed consent of participation into the study is given by the participant and his/her parent or guardian (for those aged under 18).
3. Being able to comply with the study protocol.
4. Having a DSM-5 diagnosis of depressive disorders.
5. Having a score of ≥ 40 on Children's Depression Rating Scale (CDRS-R).
6. Having a score of ≤ 41 on Horne-Östberg Morning-Eveningness Questionnaire (MEQ; classified as evening chronotype).
7. Having a sleep onset time of 11:15pm or later for 12 year olds, 11:30pm or later for 13-14 year olds, and 12:00pm or later for 15-20 years at least 3 nights per week in the past 3 months.

Exclusion Criteria:

1. A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, neurodevelopmental disorders, organic mental disorders, or intellectual disabilities.
2. Initiation of and change of medication that may interfere with circadian rhythm within past 3 months (e.g., lithium, exogenous melatonin, melatonergic antidepressants).
3. In the opinion of the research clinician, having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt).
4. Having been enrolled in any other clinical trial investigational products within one month at the entry of the study.
5. Initiation of or change in antidepressant medication within past 3 months.
6. Having been or is currently receiving any structured psychotherapy.
7. With hearing or speech deficit.
8. Night shift worker.
9. Trans-meridian flight in the past 1 month and during intervention.
10. Presence of an eye disease (e.g., retinal blindness, severe cataract, glaucoma).

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in Assessor-rated Depressive Symptoms | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Children's Depression Rating Scale (CDRS-R) is a 17-item rating scale based on a semi-structured interview with children. Possible scores range from 17 to 113, with higher scores indicating severer depressive symptoms.

SECONDARY OUTCOMES:
Change of Self-report Depressive Symptoms | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Beck's Depression Inventory (BDI-II) is a 21-item self-report rating scale measuring depression symptoms. Possible scores range from 0 to 62, with higher scores indicating more severe depressive symptoms.
Change of Suicidal Ideation | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  The Beck's Suicide Ideation Scale (BSSI) is a 19-item self-report rating scale measuring suicide ideation. Possible scores range from 0 to 38, with higher scores indicating higher suicide intention.
Change in Self-Report Chronotype Measures | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Munich Chronotype Questionnaire (MCTQ) is a self-report measures of sleeping patterns during weekdays and weekends separately. The Mid-Sleep Time (MSF/MSFsc) are used to as an indicator of chronotype, where individuals with earlier mid-sleep time reflect a morning chronotype and later mid-sleep time reflect an evening chronotype.
Change in Self-Report Circadian Typology | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  The Morningness-Eveningness Questionnaire (MEQ) is a 19-item self-report rating scale measuring circadian preference (typology). Possible scores range from 16 to 89, with lower scores indicating preference towards eveningness. Based on the conventional cut off, having a MEQ score of 16-41 is considered eveningness.
Change in Insomnia Symptoms | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Insomnia Severity Index (ISI) is a 5-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.
Change in Sleep Quality | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale consisting of 19 questions. All items are combined to form seven component scores on different aspects of sleep quality, each of which ranges from 0 to 3 points with higher scores representing more sleep disturbance. The seven component scores are added to one global score, which ranges from 0 to 21, with higher scores indicating more difficulties with sleep.
Change in Total Sleep Time (TST) measured by sleep diary | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Daily sleep diary for seven consecutive days. Total sleep time (hours) was estimated by averaging the recorded days.
Change in Sleep Onset Latency (SOL) measured by sleep diary | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Daily sleep diary for seven consecutive days. Sleep onset latency (minutes) was estimated by averaging the recorded days.
Change in Wake After Sleep Onset (WASO) measured by sleep diary | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Daily sleep diary for seven consecutive days. Wake after sleep onset (minutes) was estimated by averaging the recorded days.
Change in Sleep Efficiency (SE) measured by sleep diary | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Daily sleep diary for seven consecutive days. Sleep efficiency (in percentage, calculated by total sleep time divided by total time in bed) was estimated by averaging the recorded days.
Change in Total Sleep Time (TST) measured by actigraphy | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Actigraphy assessment for seven consecutive days. Total sleep time (hours) was estimated by averaging the recorded days.
Change in Sleep Onset Latency (SOL) measured by actigraphy | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Actigraphy assessment for seven consecutive days. Sleep onset latency (minutes) was estimated by averaging the recorded days.
Change in Wake After Sleep Onset (WASO) measured by actigraphy | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Actigraphy assessment for seven consecutive days. Wake after sleep onset (minutes) was estimated by averaging the recorded days.
Change in Sleep Efficiency (SE) measured by actigraphy | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Actigraphy assessment for seven consecutive days. Sleep efficiency (in percentage, calculated by total sleep time divided by total time in bed) was estimated by averaging the recorded days.
Change in Actigraphic Circadian Measures - L5 computed by nonparametric circadian rhythm analysis | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Actigraphic assessment for seven consecutive days. The start times and average activity of L5 (i.e., five hours of least activity within a 24-hour period) is computed by the nonparametric circadian rhythm analysis.
Change in Actigraphic Circadian Measures - M10 computed by nonparametric circadian rhythm analysis | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Actigraphic assessment for seven consecutive days. The start times and average activity of M10 (i.e., 10 hours of maximal activity within a 24-hour period) is computed by the nonparametric circadian rhythm analysis.
Change in Actigraphic Circadian Measures - acrophase computed by cosinor analysis | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Actigraphic assessment for seven consecutive days. The acrophase (defined as time of maximum activity express as clock time) is computed by cosinor analysis.
Change in Actigraphic Circadian Measures - amplitude computed by cosinor analysis | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Actigraphic assessment for seven consecutive days. The amplitude (defined as the differences in distance from the peak to the nadir) is computed by cosinor analysis.
Change in Actigraphic Circadian Measures - MESOR computed by cosinor analysis | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Actigraphic assessment for seven consecutive days. The MESOR (defined as the mean activity level) is computed by cosinor analysis.
Change in Objective Physiological Circadian Measures | Baseline, one-week post-treatment/Week 9
  Home-based dim-light melatonin onset assessment (expressed as time value hh:mm) is determined by 10-hour salivary melatonin collected at 30-minute intervals.
Change in Daytime Sleepiness | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Paediatric Daytime Sleepiness Scale (PDSS) is an 8-item self-rated scale measuring daytime sleepiness, ranging in total scores from 0 to 32 with higher scores indicating more sleepiness.
Change in Daytime Fatigue | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  Multidimensional Fatigue Inventory (MFI) is a 20-item self-rated scale on fatigue symptoms. There are three subscales, measuring the physical (possibly scored from 7 to 35), mental (possibly scored from 6 to 30), and spiritual (possibly scored from 7 to 35), dimensions of fatigue. A grand total score can be calculated by summing up the three sub scores. In all cases, a higher score represents higher fatigue symptoms.
Change in Quality of Life | Baseline and one-week post-treatment/Week 9 for all participants, and post-treatment 1-month follow-up and post-treatment 6-month follow-up for the participants in the treatment groups
  KIDSCREEN-27 is a 27-item self-rated scale measuring health related quality of life measure for children and adolescents. There are five subscales on: physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong